CLINICAL TRIAL: NCT04942769
Title: Study on the Effect of Selenium Supplementation on the Structure and Function of Autoimmune Thyroiditis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Professor and Director, Department of Endocrinology, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-310
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Selenium
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Intervention Model Description: patients with Autoimmune thyroiditis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- selenium (Experimental): selenium was administered to patients with autoimmune thyroiditis
  Interventions: Drug: Selenium

INTERVENTIONS:
Drug: Selenium — selenium 100ug ，take it orally twice daily

SUMMARY:
To evaluate the effects of exogenous selenium supplementation on autoimmune thyroiditis.

DETAILED DESCRIPTION:
In patients with autoimmune thyroiditis， investigators compared changes in thyroid function, anti-thyroid peroxidase antibody, anti-thyroglobulin antibody, thyroid magnetic resonance T1-mapping values and metabolic indicatorsfrom baseline to the end of treatment (12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 75
* Clinical diagnosis of autoimmune thyroiditis, serum TPOAb and TGAB positive
* Thyroid function is normal, and no drugs affecting thyroid function such as Umetole and Serge have been used

Exclusion Criteria:

* The contraindications indicated in the Chinese instructions of the drug
* Hypothyroidism, hyperthyroidism
* Liver function impairment
* Renal function impairment
* Claustrophobia
* Mental disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
anti-thyroglobulin antibody changes | Changes from baseline and 3 months during follow-up
  Changes from baseline and 3 months during follow-up
T1-mapping values of Thyroid MRI | Changes from baseline and 3 months during follow-up
  Changes from baseline and 3 months during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China